CLINICAL TRIAL: NCT04144296
Title: Mathematical Arterialisation of Capillary Blood for Blood Gas Analysis in Critical Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Collaborators: OBI Medical (Unknown)
Responsible Party: Principal Investigator, PD Dr. Tobias Müller, Consultant, RWTH Aachen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-125
Record Dates: First submitted 2019-10-21; First posted 2019-10-30 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Lung Diseases
Keywords: Arterial blood gas analysis; Capillary blood gas analysis
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Other): All patient will be included in this arm
  Interventions: Diagnostic Test: Study procedure

INTERVENTIONS:
Diagnostic Test: Study procedure — * Measurement of the flow rate of supplemental oxygen
  * Measurement of the peripheral arterial saturation (SpO2) by pulse oximetry
  * Taking of an ABG sample (ABG1) from the arterial line
  * Taking of capillary blood gas analysis from the earlobe and from the finger tip
  * Taking of an a second ABG (ABG2) from the arterial line

SUMMARY:
The aim of the study is to compare capillary blood gas analysis compensated by v-TAC software (aCBGE, aCBGF) to arterial blood gas analysis (ABG) in terms of pH, pCO2 and pO2 and the clinical usefulness of this method compared to the gold standard of ABG.

DETAILED DESCRIPTION:
In clinical practice blood gas analysis is an essential tool for monitoring respiratory status. The gold-standard method is arterial blood gas analysis (ABG) of blood from the patient's radial or femoral artery. An alternative to arterial sampling commonly used is arterialized capillary blood gas analysis from the earlobe (CBGE). Though CBGE is less invasive and can be performed by non-medical staff, it is less useful in the acute setting because an adequate vasodilatation is needed which typically lasts for at least 10 minutes and the quality of results tends to be operator dependable. Different trials have evaluated the agreement between ABG and CBGE. Whereas a close agreement between ABG and CBGE has been found for evaluating pH and the partial pressure of carbon dioxide (PCO2), several trials showed considerable variations for the partial pressure of oxygen (PO2) and that CBGE tends to underestimate PO2. Similar findings apply for capillary blood gas analysis from the fingertip (CBGF) which is even less accurate compared to CBGE in estimating PO2. Recently a method has been developed to calculate ABG values mathematically from peripheral venous blood, supplemented with oxygen saturation (SpO2) measurement by pulse oximetry, by use of venous-to-arterial conversion (v-TAC) software (OBI Medical, Denmark). The principle of the method is a mathematical transformation of venous blood gas analysis (VBG) values to arterialised values (aVBG) by simulating the transport of blood back through the tissue (6). This approach leads to a clinically acceptable agreement between ABG and aVBG for pH and PCO2. For PO2 the limits of agreement of aVBG are similar to those of PO2 from CBGE for values below 75 mmHg and with mean bias close to zero. However, it has not been evaluated previously whether v-TAC software can be used to calculate ABG values from CBGE (aCBGE) or CBGF (aCBGF). As CBGE and CBGF values are much closer to ABG values, compared to VBG values, the agreement between aCBGE/aCBGF and ABG in terms of pH, PCO2 and pO2 might be better compared to CBG without mathematical arterialisation by v-TAC.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the intensive / intermediate care or weaning unit at the department of pneumology and intensive care medicine of the university hospital RWTH Aachen
* Arterial line inserted to monitor the patient's blood pressure or respiratory status
* Male or female aged ≥ 18 years
* Written informed consent prior to study participation
* The subject is willing and able to follow the procedures outlined in the protocol

Exclusion Criteria:

* Hemodynamic instability
* Impaired perfusion of peripheral limbs e.g. due to severe heart failure
* Pregnant and lactating females. Pregnancy will be ruled out in females of childbearing age by pregnancy test.
* Patient has been committed to an institution by legal or regulatory order
* The subject is mentally or legally incapacitated

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of pO2 Levels (in mmHg) in capillary blood samples corrected with VTAC Software to arterial blood samples | 10 minutes after the first blood sample is taken
  Capillary and arterial pO2 Levels will be measured using a blood gas analyser. Afterwards pO2 levels in the capillary sample will be compensated by VTAC software and compensated pO2 levels will be compared to arterial PO2 levels using the Bland-Altman method.

SECONDARY OUTCOMES:
Comparison of pCO2 Levels (in mmHg) in capillary blood samples corrected with VTAC Software to arterial blood samples | 10 minutes after the first blood sample is taken
  Capillary and arterial pCO2 Levels will be measured using a blood gas analyser. Afterwards pCO2 levels in the capillary sample will be compensated by VTAC software and compensated pCO2 levels will be compared to arterial PCO2 levels using the Bland-Altman method.
Comparison of pH in capillary blood samples corrected with VTAC Software to arterial blood samples | 10 minutes after the first blood sample is taken
  Capillary and arterial pH will be measured using a blood gas analyser. Afterwards pH in the capillary sample will be compensated by VTAC software and compensated pH will be compared to arterial pH levels using the Bland-Altman method.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for pneumology and internal intensive care, Aachen, Germany